CLINICAL TRIAL: NCT04449770
Title: A Study on the Use of an Established Novel Height-based Formula for Predicting the Insertion Depth of Left-sided Double and the Role of Fiberoptic Bronchoscopy
Brief Title: Height-based Formula for Predicting the Insertion Depth of Left-sided Double and the Role of Fiberoptic Bronchoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, A.Eldawlatly, professor, King Saud University
Other Study IDs: E-18-3064/IRB 06.05.2018
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Thoracic Anesthesia
Keywords: Thoracic anesthesia; Double lumen tube; Height based formula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: double lumen tube — prospective cohort study

SUMMARY:
The use of height based formula to predict insertion depth of left-sided double lumen tube in thoracic surgery is now well established. The investigators have developed a formula to be used and published recently. The investigators verified the formula with the use of FOB. This observational study we are going to use with FOB checking if needed.

DETAILED DESCRIPTION:
The use of a height-based formula to predict the insertion depth of left-sided double-lumen tubes in thoracic surgery is now well established. The investigators have developed a formula to be used and published recently. The investigators verified the formula with the use of FOB. This observational study will use FOB checking if needed.

Our hypothesis is that DLT can insert without the use of FOB in most of the cases. That doesn't mean FOB is less required.

ELIGIBILITY:
Inclusion Criteria:

* patients whose procedure required placement of an LDLT

Exclusion Criteria:

* patients with intraluminal bronchial lesions and patients with a difficult airway.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult patients aged 20-60 yr undergoing thoracic surgery with the use of left-sided DLT for lung isolation
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
correct position of DLT with proper lung deflation without use of FOB | during surgical time
  proper lung deflation, surgeon satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided